CLINICAL TRIAL: NCT03225261
Title: The Effect of Citrus Extract Administration on Gastrointestinal Health
Brief Title: The Effect of Citrus Extract on Gastrointestinal Health
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Yala Stevens, MSc., Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 173003
Record Dates: First submitted 2017-06-09; First posted 2017-07-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — grapefruit seed extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citrus extract (Experimental): Citrus extract
  Interventions: Dietary Supplement: Citrus extract
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Citrus extract — Citrus extract
  Arms: Citrus extract
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
This randomized, parallel, double-blind, placebo-controlled trial aims to determine the effects of daily administration of citrus extract over a period of 8 weeks on gastrointestinal health in patients with irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IBS
* Calprotectin levels 15-150 µg/g feces
* Age 18-70 years
* BMI < 35 kg/m2

Exclusion Criteria:

* Comorbidities that may influence gut microbiota composition or which might limit participation in or completion of the study protocol (to be decided by the principle investigator)
* Abdominal surgery interfering with gastrointestinal function (to be decided by the principle investigator)
* Use of immunosuppressive drugs within 3 months before study period
* Use of other medication interfering with endpoints
* Changes in medication that may significantly affect the study outcome according to the investigator's judgment within 1 month prior to the study
* Changes in clinical activity scores within 3 weeks prior to the study
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator) in the 180 days prior to the study
* Use of dietary supplements containing antioxidants, minerals and vitamins
* Excessive intake of foods with a high polyphenol concentration
* Use of antibiotics within 3 months prior to the start of study
* Use of pre-or probiotics within 1 month prior to the study
* Use of oral corticosteroids within 1 month prior to the study
* Blood donation within 1 month prior to the study
* Known pregnancy or lactation.
* Excessive drinking (>20 alcoholic consumptions per week)
* History of any side effects towards the intake of flavonoids or citrus fruits

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-13 (Actual)

PRIMARY OUTCOMES:
The effect on intestinal inflammation, measured by fecal calprotectin levels. | 8 weeks
  The primary objective is to assess the effect of 500 mg citrus extract on intestinal flammation after 8 weeks of administration, by measuring fecal calprotectin in IBS patients with moderately increased fecal calprotectin levels.

SECONDARY OUTCOMES:
The effect on microbial metabolic activity, measured by fecal short chain fatty acids (SCFA). | 8 weeks
The effect on fecal microbiota composition, assessed by next generation sequencing. | 8 weeks
The effect on fecal microbiota functional capacity, assessed by next generation sequencing. | 8 weeks
The effect on the systemic immune response, measured by cytokine production capacity of stimulated whole blood | 8 weeks
The effect on disease symptoms, measured by patient reported outcomes (GSRS). | 8 weeks
The effect on disease symptoms, measured by patient reported outcomes (symptom diary). | 8 weeks
The effect on stool frequency, measured by Bristol Stool Chart. | 8 weeks
The effect on stool consistency, measured by Bristol Stool Chart. | 8 weeks
The effect on blood markers for oxidative stress, measured by MDA concentration in blood. | 8 weeks
The effect on blood markers for antioxidant capacity, measured by blood total antioxidant capacity. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ad Masclee, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No